CLINICAL TRIAL: NCT03680781
Title: Accelerated Theta Burst in Treatment-Resistant Depression: A Dose Finding and Biomarker Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gregory Sahlem, Clinical Assistant Professor, Department of Psychiatry & Behavioral Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-44150
Record Dates: First submitted 2018-09-10; First posted 2018-09-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Accelerated theta burst treatment (Experimental): All participants will receive theta-burst TMS.
  Interventions: Device: Intermittent theta-burst stimulation (iTBS)

INTERVENTIONS:
Device: Intermittent theta-burst stimulation (iTBS) — Participants will receive iTBS to the left DLPFC or bilateral DLPFC, to the right and left DLPFC. The DLPFC will be targeted utilizing either Localite's neuronavigation system or Nexstim's eField neuronavigation system. Stimulation intensity will be standardized at 90% of RMT and adjusted to the skull to cortical surface distance (see Nahas 2004).
  Stimulation will be delivered to the L-DLPFC or bilateral DLPFC using either a MagVenture MagPro X100 or a Nexstim TMS device.

SUMMARY:
This study evaluates the effectiveness of re-treatment using accelerated schedule of intermittent theta-burst stimulation for treatment-resistant depression. This is an open label study.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established technology as therapy for treatment-resistant depression. The approved method for treatment is 10Hz stimulation for 40 min over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been very successful. The limitations of this approach include the duration of the treatment (approximately 40 minutes per treatment session). Recently, researchers have aggressively pursued modifying the treatment parameters to reduce treatment times with some preliminary success. This study will investigate the efficacy of a further modified protocol, creating a more rapid form of the treatment and look at the change in neuroimaging biomarkers. In particular, this study will determine the efficacy of re-treatment in individuals who have already experienced benefit of the accelerated protocol to ensure results can be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age.
* Able to provide informed consent.
* Diagnosed with Major Depressive Disorder (MDD) or bipolar affective disorder 2 and currently experiencing a Major Depressive Episode (MDE).
* prior exposure to rTMS
* Participants must qualify as "moderate or severe treatment refractory" using the Maudsley staging method.
* Participants may continue antidepressant regimen, but must be stable for 6 weeks prior to enrollment in the study. They must maintain that same antidepressant regimen throughout the study duration.
* Participants are required to have a stable psychiatrist for the duration of study enrollment.

Exclusion Criteria:

* History of MI, CABG, CHF, or other cardiac history
* Any neurological conditions
* History of epilepsy
* OCD
* Independent sleep disorder
* Autism Spectrum Disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage change in Hamilton Depression Rating Scale 21-Item score | Difference between baseline and one month after aiTBS treatment
  A 21 item clinical assessment tool used to rate a patient's level of depression - total scores range from 0-63 with higher scores indicating worse depression

SECONDARY OUTCOMES:
Change in Hamilton Rating Scale for Depression (HAMD-17) | Pretreatment, immediately posttreatment, 2 weeks posttreatment, 4 weeks posttreatment
  A provider administered questionnaire used to rate a patient's level of depression - total scores range from 0-52 with higher scores indicating worse depression
Change in The Scale for Suicide Ideation | Pretreatment, immediately posttreatment, 2 weeks posttreatment, 4 weeks posttreatment
  A rating scale that measures the current intensity of specific attitudes, behaviors, and plans to commit suicide - total scores range from 0-38 with higher scores indicating greater suicidality
Change in Hamilton Rating Scale for Depression (HAMD-6) | Every day of stimulation, follow-up every 2 weeks after treatment for 6 months by telephone]
  rate a patient's level of depression - total scores range from 0-22 with higher scores indicating worse depression
Change from baseline functional connectivity | Pretreatment, immediately post-treatment, 4 weeks post-treatment
  We will assess functional connectivity as seen on resting state fMRI, between the subcallosal cingulate to the default mode network and within the default mode network.
Change in Beck Depression Inventory (BDI) | Pretreatment, immediately post-treatment, 4 weeks post-treatment
  Self-report measure of depressive symptoms - total scores range from 0-63 with higher scores indicating worse depression
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) | Pretreatment, immediately post-treatment, 4 weeks post-treatment
  A 10 item clinician rated measure of depressive symptoms - total scores range from 0-60 with higher scores indicating worse depression

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, MD, Principal Investigator — Stanford University
Locations (1):
- Department of Psychiatry and Behavioral Sciences, Stanford School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Jelic MB, Milanovic SD, Filipovic SR. Differential effects of facilitatory and inhibitory theta burst stimulation of the primary motor cortex on motor learning. Clin Neurophysiol. 2015 May;126(5):1016-23. doi: 10.1016/j.clinph.2014.09.003. Epub 2014 Sep 16. PMID 25281475
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537